CLINICAL TRIAL: NCT03326050
Title: Gemifloxacin Versus Ciprofloxacin Versus Rifampicin in Treatment of Rhinoscleroma
Brief Title: Comparison Between Rifampicin and Gemifloxacin and Ciprofloxacin in Treatment of Rhinoscleroma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, asmaa ahmed bekheit, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rhinoscleroma
Record Dates: First submitted 2017-10-18; First posted 2017-10-30 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Rhinoscleroma
Keywords: Rhinoscleroma; Gemifloxacin; Ciprofloxacin
MeSH Terms: conditions — Rhinoscleroma | interventions — Gemifloxacin; Tablets; Ciprofloxacin; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- gemifloxacin and Rifampicin (Placebo Comparator): first group will be given a short course (four weeks) of oral Gemifloxacin 320 mg once dailygroup will be given the usual regimen given for free by the Ministry of Health in Egypt; Rifampicin 300 mg twice daily for three months..
  Interventions: Drug: Gemifloxacin; Drug: Ciprofloxacin; Drug: Rifampicin
- gemifloxacin and ciprofloxacin (Placebo Comparator): . group will be given a short course (four weeks) of oral Gemifloxacin 320 mg once daily group will be given a short course (four weeks) of oral Ciprofloxacin 750 mg twice daily
  Interventions: Drug: Gemifloxacin; Drug: Ciprofloxacin; Drug: Rifampicin
- gemifloxacin and placipo (Placebo Comparator): .group will be given a short course (four weeks) of oral Gemifloxacin 320 mg once daily
  Interventions: Drug: Gemifloxacin; Drug: Ciprofloxacin; Drug: Rifampicin

INTERVENTIONS:
Drug: Gemifloxacin — Gemifloxacin 320Mg Oral Tablet once daily
  Other Names: Gemifloxacin 320Mg Oral Tablet
Drug: Ciprofloxacin — cipro 750 tablet twice daily
  Other Names: Cipro 750Mg Tablet
Drug: Rifampicin — Rifampicin 150Mg Capsule twice daily
  Other Names: Rifampicin 150Mg Capsule

SUMMARY:
gemifloxacin versus ciprofloxacin and rifampicin in treatment of rhinoscleroma

DETAILED DESCRIPTION:
Rhinoscleroma is a chronic specific granulomatous inflammation affecting nose in 95-100% but can affect any part of respiratory tract.(1)

It is an endemic disease in Egypt. It is endemic as well in sporadic areas worldwide including Central America, Chili, Central Africa, India, Indonesia and Middle East countries.(2) It is completely eradicated from the developed communities.

If not treated early, the disease progresses to the final sclerotic phase where permanent complications including nasal deformities, anosmia, dysphonia, dysphagia and stridor could happen.(3-5)

Of the wide treatments range (antibiotic combinations, cytostatic drugs, radiation, and laser), none is ideal. The causative organism is resistant to most antibiotics and, being intracellular, is not always exposed to sufficient concentrations of drug. A clinical cure is hard to identify because the end-stage is mucosal fibrosis which, even without active infection, interferes with normal function of the upper respiratory tract. The fibrosed mucosa, especially in crusts, can become secondarily infected with bacteria, which may include klebsiella.(6)

Rifampin (7), streptomycin (8), ciprofloxacin (5) and levofloxacin (9) have been used in treatment of rhinoscleroma.

Most patients are from a low socioeconomic group and cannot afford the price of antibiotics to which klebsiella is susceptible. (6)

The usual regimen given for free by the Ministry of Health in Egypt in histologically positive cases is Rifampicin 300 mg twice daily for six months (based on a nasal biopsy and documented as a Tuberculosis, not rhinoscleroma, to allow free delivery of the medication) then another biopsy is taken to identify if cure or not. If not, Rifampicin is given for another six months and so on.

Unfortunately, due to the high level of antimicrobial resistance, poor patients' compliance, and drugs side effects, the treatment failure rate is increasing. So there is a real need for an alternative drug that is effective, safe and has a short treatment course.

Gemifloxacin is a new fluoroquinolone that has bactericidal activity. It has good intracellular penetration and low toxicity.(10) It is more potent than ciprofloxacin, ofloxacin and levofloxacin.(11)

ELIGIBILITY:
Inclusion Criteria:

1. Age above 18 years
2. Active rhinoscleroma proved both clinically and histopathologically

Exclusion Criteria:

1. Patients younger than 18 years old.
2. inactive Rhinoscleroma
3. Contraindication to treatment severe renal or hepatic impairment
4. Refusal of enrollment in the research by the patient

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-02 (Estimated); Primary Completion 2018-09-01 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
clinical examination., nasal crustation, | monthly evaluation for 6 months
  nasal crusting, O= no symptoms, 1 = present monthly 2= present weekly, 3 = present daily, 4 = always present, and 5 = incapacitating). (6)
clinical examination purulent secretions | monthly evaluation for 6 months
  purulent secretions (O= no symptoms, 1 = present monthly 2= present weekly, 3 = present daily, 4 = always present, and 5 = incapacitating). (6)
• Full ENT history | monthly evaluation for 6 months
  purulent rhinorrhea, postnasal discharge, nasal crustation, hyposmia, and nasal obstruction

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed mohamed, lecturer, Study Director — assiut yunveristy
Locations (1):
- Asmaa Ahmed, Asyut, Egypt

REFERENCES:
- [Result] Ahmed AR, El-Badawy ZH, Mohamed IR, Abdelhameed WA. Rhinoscleroma: a detailed histopathological diagnostic insight. Int J Clin Exp Pathol. 2015 Jul 1;8(7):8438-45. eCollection 2015. PMID 26339415
- [Result] The Editors. Rhinoscleroma. J Med Microbiol. 2000 May;49(5):395-396. doi: 10.1099/0022-1317-49-5-395. No abstract available. PMID 10798549
- [Result] Zhong Q, Guo W, Chen X, Ni X, Fang J, Huang Z, Zhang S. Rhinoscleroma: a retrospective study of pathologic and clinical features. J Otolaryngol Head Neck Surg. 2011 Apr;40(2):167-74. PMID 21453653
- [Result] Fawaz S, Tiba M, Salman M, Othman H. Clinical, radiological and pathological study of 88 cases of typical and complicated scleroma. Clin Respir J. 2011 Apr;5(2):112-21. doi: 10.1111/j.1752-699X.2010.00207.x. PMID 21410904
- [Result] Bailhache A, Dehesdin D, Francois A, Marie JP, Choussy O. Rhinoscleroma of the sinuses. Rhinology. 2008 Dec;46(4):338-41. PMID 19146007
- [Result] Borgstein J, Sada E, Cortes R. Ciprofloxacin for rhinoscleroma and ozena. Lancet. 1993 Jul 10;342(8863):122. doi: 10.1016/0140-6736(93)91329-k. No abstract available. PMID 8100894
- [Result] Gamea AM, el-Tatawi FA. The effect of rifampicin on rhinoscleroma: an electron microscopic study. J Laryngol Otol. 1990 Oct;104(10):772-7. doi: 10.1017/s002221510011388x. PMID 2246576
- [Result] Toppozada HH, Gaafar HA. The effect of streptomycin and irradiation on rhinoscleroma (electron microscopic study). J Laryngol Otol. 1986 Jul;100(7):809-15. doi: 10.1017/s0022215100100118. PMID 3734600
- [Result] Pound MW, Fulton KB, Chima CO. Successful treatment of Klebsiella rhinoscleromatis bacteremia with levofloxacin. Pharmacotherapy. 2007 Jan;27(1):161-3. doi: 10.1592/phco.27.1.161. PMID 17192170
- [Result] Saravolatz LD, Leggett J. Gatifloxacin, gemifloxacin, and moxifloxacin: the role of 3 newer fluoroquinolones. Clin Infect Dis. 2003 Nov 1;37(9):1210-5. doi: 10.1086/378809. Epub 2003 Oct 2. PMID 14557966
- [Result] Hoban DJ, Bouchillon SK, Johnson JL, Zhanel GG, Butler DL, Miller LA, Poupard JA; Gemifloxacin Surveillance Study Research Group. Comparative in vitro activity of gemifloxacin, ciprofloxacin, levofloxacin and ofloxacin in a North American surveillance study. Diagn Microbiol Infect Dis. 2001 May-Jun;40(1-2):51-7. doi: 10.1016/s0732-8893(01)00241-3. PMID 11448564